CLINICAL TRIAL: NCT05608902
Title: Structural Description of Skin Biopsies With Dynamic Full-field Optical Coherence Tomography on Suspected Basal Cell Carcinoma Lesions, a Pilot Study
Brief Title: Structural Description of Skin Biopsies With Dynamic Full-field Optical Coherence Tomography on Suspected Basal Cell Carcinoma Lesions, a Pilot Study (DOCTOBA)
Acronym: DOCTOBA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Responsible Party: Principal Investigator, Thomas Maldiney, Doctor, Centre Hospitalier William Morey - Chalon sur Saône
Other Study IDs: DermatOCT1
Record Dates: First submitted 2022-10-21; First posted 2022-11-08 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Basal Cell Carcinoma; Tomography, Optical Coherence
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DOCTOBA cohort: Patients > 18 years of age with suspected basal cell carcinoma requiring biopsy or skin resection in the dermatology department
  Interventions: Other: Dynamic full-field optical coherence tomography analysis of skin biopsy or resection

INTERVENTIONS:
Other: Dynamic full-field optical coherence tomography analysis of skin biopsy or resection — Dynamic full-field optical coherence tomography analysis of skin biopsy or resection in the dermatology department before conventional histopathological analysis

SUMMARY:
Basal cell carcinoma (BCC) are the most frequent skin cancers. Their incidence is constantly increasing. BCC diagnosis is first clinically suspected and then confirmed following histological examination of either a skin biopsy or the excisional specimen. Surgery is the first-line treatment and some procedures (notably Mohs surgery) require extemporaneous histological analysis of the edges to ensure a complete excision. Such on-site histopathological examination can be time consuming and associated with decreased sensitivity. Skin imaging techniques have already been tested to overcome these limitations and seem promising. Although some of them - such as confocal microscopy - are already even used in vivo, there is to date no report of the use of full-field optical coherence tomography for the diagnosis of BCC.

The DOCTOBA study intends to describe direct histopathological examination of fresh skin biopsy or excisional specimen with dynamic full-field optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

- patient > 18 years of age who received skin biopsy or excision of basal cell carcinoma suspected lesion between start study date and primary completion date

Exclusion Criteria:

* inability to perform dynamic full-field optical coherence tomography observation at the moment of skin biopsy
* diagnosis of basal cell carcinoma disproved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient > 18 years of age who received skin biopsy or excision of basal cell carcinoma suspected lesion
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Histopathological analysis of basal cell carcinoma with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following skin biopsy or resection
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify and characterize the usual basal cell carcinoma, comprising basaloid cells with a thin pale cytoplasm surrounding round or oval nuclei with a rough granulated chromatin pattern, palisade arrangement, artificially created slits, rather chaotic internal arrangement, mitoses and necrosis ; but also to identify the different sub-types of basal cell carcinoma (nodular, superficial, infiltrating, scleroderma).

SECONDARY OUTCOMES:
Histopathological analysis of healthy skin with dynamic full-field optical coherence tomography | Outcome measure is assessed 15 days following skin biopsy or resection
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify the normal structures of the skin (meaning not affected by carcinoma), i.e. the different layers of the skin (epidermis, dermis and subcutaneous tissue) and the skin appendages (hair follicles and glands), also to recognize the different cells and components (keratinocytes, melanocytes, Langerhans cells, Merkel celles and collagen) and underlayers (stratum corneum, stratum granulosum, stratum spinosum, stratum basale, epidermal cretes, dermo-hypodermic junction, papillary dermis and reticularis dermis).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Maldiney, Principal Investigator — Centre Hospitalier William Morey - Chalon sur Saône
Locations (1):
- Centre Hospitalier William Morey - Chalon sur Saône, Chalon-sur-Saône, Saône-et-Loire, France

IPD SHARING:
Plan to Share IPD: Undecided